CLINICAL TRIAL: NCT07299708
Title: Effects of Sleep Quality, Anxiety, and Digital Behavior on Labor Progression in Term Primiparous Women: A Prospective Observational Study
Acronym: SAD-LABOR
Status: Completed | Type: Observational
Sponsor: Tepecik Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Fatih Yıldırım, Obstetrics and Gynecology Specialist, Principal Investigator, Tepecik Training and Research Hospital
Other Study IDs: TEPECIK-SAD-LABOR; TEPECIK-EC-2025-07-10 (06/08/2 (Registry Identifier: İzmir Tepecik Training and Research Hospital Ethics Committee)
Record Dates: First submitted 2025-11-23; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Labor Progression; Pregnancy
Keywords: Sleep Quality; Anxiety; Digital Behavior; Primiparous Women; Childbirth; Oxytocin Augmentation
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Primiparous Cohort: Term primiparous women assessed for sleep quality, anxiety, digital behavior, and followed through spontaneous labor.
  Interventions: Other: No Intervention: Observational Cohort

INTERVENTIONS:
Other: No Intervention: Observational Cohort — Observational study with no assigned treatment or intervention.

SUMMARY:
This prospective observational study evaluates whether maternal sleep quality, anxiety levels, and nighttime digital behavior are associated with labor progression among term primiparous women. Sleep quality and anxiety are assessed before the onset of labor during routine antenatal visits using validated instruments, including the Pittsburgh Sleep Quality Index (PSQI) and the Beck Anxiety Inventory (BAI). Nighttime digital behavior characteristics, such as screen exposure and smartphone use prior to sleep, are recorded through standardized antenatal interviews.

Labor outcomes, including the duration of the latent, active, and second stages of labor, requirement for oxytocin augmentation, use of analgesia, and mode of delivery, are prospectively documented from hospital admission until birth. By examining behavioral and psychological factors prior to labor onset, the study aims to determine whether poor sleep quality, increased anxiety, or irregular nighttime digital activity are associated with prolonged labor phases or greater need for obstetric interventions.

DETAILED DESCRIPTION:
This prospective observational cohort study investigates the influence of maternal sleep quality, anxiety levels, and nighttime digital device use on labor progression among term primiparous women. Eligible participants were term primiparous women attending routine antenatal follow-up at Izmir Tepecik Training and Research Hospital. All psychosocial assessments were completed prior to the onset of labor. Sleep quality was evaluated using the Pittsburgh Sleep Quality Index (PSQI), and anxiety levels were assessed using the Beck Anxiety Inventory (BAI). Nighttime digital behavior characteristics were documented through structured antenatal interviews and included pre-sleep screen exposure, smartphone use in bed, frequency of nighttime phone checking, and the type of digital content viewed before sleep.

Participants were subsequently followed through spontaneous labor, and labor-related data were collected prospectively. Initial labor characteristics documented at hospital admission included cervical dilation, contraction pattern, and overall clinical presentation. Additional labor outcomes, including the duration of the latent, active, and second stages of labor, use of oxytocin augmentation, requirement for epidural or opioid analgesia, operative vaginal delivery, cesarean delivery, and neonatal outcomes, were recorded systematically according to standardized institutional protocols.

The primary aim of the study is to determine whether poor sleep quality, elevated anxiety levels, or increased nighttime digital device use are associated with prolonged labor or dysfunctional labor patterns. Secondary aims include examining whether interactions between digital behavior variables and psychological factors contribute to variations in maternal labor physiology or to increased obstetric intervention rates.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women at ≥ 37 weeks of gestation
* Completion of PSQI (sleep quality) and BAI (anxiety) assessments during antenatal clinic visit
* Singleton pregnancy
* Cephalic presentation
* Age 18 to 50 years
* Planning to deliver at the study hospital
* Able to provide informed consent

Exclusion Criteria:

* Multiple pregnancy
* Non-cephalic presentation
* Delivery occurring at another hospital or birth center
* Elective planned cesarean delivery
* Major fetal anomaly
* Placenta previa or placenta accreta spectrum
* Preeclampsia, eclampsia, HELLP syndrome
* Gestational diabetes requiring insulin
* Chronic medical disorders affecting labor physiology
* Use of sedative, hypnotic, or psychotropic medications
* Inability to complete questionnaires

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only self-identified women who are biologically female and pregnant are eligible to participate in this study.
Study Population: This study population consists of term primiparous pregnant women who attended routine antenatal follow-up at Izmir Tepecik Training and Research Hospital and subsequently experienced spontaneous onset of labor. All participants were healthy, low-risk obstetric patients with singleton, cephalic presentations and no medical or obstetric complications.
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2025-08-10 (Actual); Primary Completion 2025-11-25 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Duration of Active Labor | From onset of active labor (≥4 cm) until full cervical dilatation (10 cm), typically within 2 to 12 hours.
  Time in minutes from the onset of active labor (defined as cervical dilatation of ≥4 cm with regular contractions) to full cervical dilatation (10 cm). Data will be obtained prospectively from electronic delivery records.

SECONDARY OUTCOMES:
Duration of Latent Phase of Labor | From onset of regular contractions until onset of active labor (≥4 cm), typically lasting up to 20 hours.
  Time (in minutes) from onset of regular contractions to 4 cm cervical dilation, recorded prospectively from labor charts. Evaluated in relation to sleep quality, anxiety levels, and nighttime digital behavior.
Duration of Second Stage of Labor | From full dilatation (10 cm) until birth, typically lasting up to 3 hours.
  Time in minutes from full cervical dilatation (10 cm) to the delivery of the neonate. Pushing time will be recorded prospectively.
Oxytocin Augmentation Requirement | From admission in active labor (≥4 cm) until delivery, typically within 2 to 12 hours.
  Proportion of participants requiring oxytocin infusion due to inadequate uterine contractions or labor arrest, as documented by obstetric staff.
Mode of Delivery | Assessed at delivery.
  Rates of spontaneous vaginal delivery, operative vaginal delivery, and cesarean delivery, evaluated according to sleep, anxiety, and digital behavior parameters.
Use of Epidural Analgesia | From onset of active labor (≥4 cm) until delivery, typically within 2 to 12 hours.
  Proportion of participants receiving epidural anesthesia for labor pain management, and its association with sleep quality, anxiety scores, and digital device use.
APGAR Score at 1 and 5 Minutes | Assessed at 1 and 5 minutes after birth.
  Apgar scores assessed at 1 and 5 minutes after birth.
Neonatal Intensive Care Unit (NICU) Admission | Assessed within the first 24 hours after birth.
  Number of neonates requiring admission to the neonatal intensive care unit.
Birth Weight | Assessed at birth.
  Neonatal birth weight measured in grams immediately after delivery.

CONTACTS AND LOCATIONS:
Locations (1):
- Tepecik Training and Research Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared. The dataset contains sensitive clinical information from pregnant women and cannot be made publicly available due to institutional and national data protection regulations. Summary results will be published in peer-reviewed journals, but no individual-level data will be released.